CLINICAL TRIAL: NCT01909414
Title: A Phase 1 Study of the Safety and Immunogenicity of DNA/MVA Immunizations With Co-Expressed GM-CSF in HIV-1 Infected Young Adults With Suppressed Viremia on HAART
Brief Title: Evaluating the Safety and Immune Response of DNA/MVA Vaccines in HIV-1-Infected Young Adults Taking Anti-HIV Medications
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P1082; 10776 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2013-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Arm A: GEO-D03 DNA and MVA/HIV62B vaccines (Experimental): At study entry and Week 8, participants will receive the GEO-D03 DNA vaccine administered as 1 mL intramuscularly (IM) in either deltoid. At Weeks 16 and 24, they will receive the MVA/HIV62B vaccine administered as 1 mL IM in either deltoid.
  Interventions: Biological: GEO-D03 DNA Vaccine; Biological: MVA/HIV62B Vaccine
- Arm B: Placebo for GEO-D03 and MVA/HIV62B (Placebo Comparator): At study entry and Week 8, participants will receive the placebo for GEO-D03 DNA vaccine administered as 1 mL IM in either deltoid. At Weeks 16 and 24, they will receive the placebo for MVA/HIV62B vaccine administered as 1 mL IM in either deltoid.
  Interventions: Biological: Placebo for DNA GEO-D03; Biological: Placebo for MVA/HIV62B Vaccine

INTERVENTIONS:
Biological: GEO-D03 DNA Vaccine — DNA GEO-D03 vaccine will be administered as a 3 mg dose IM.
  Arms: Arm A: GEO-D03 DNA and MVA/HIV62B vaccines
Biological: MVA/HIV62B Vaccine — MVA/HIV62B vaccine will be administered as a 1 x 10^8 TCID50 dose IM.
  Arms: Arm A: GEO-D03 DNA and MVA/HIV62B vaccines
Biological: Placebo for DNA GEO-D03 — Placebo for DNA GEO-D03 (administered as 0.9 percent Sodium Chloride for Injection) will be administered IM.
  Arms: Arm B: Placebo for GEO-D03 and MVA/HIV62B
Biological: Placebo for MVA/HIV62B Vaccine — Placebo for MVA/HIV62B 1 x 10^8 TCID50 (administered as 0.9 percent Sodium Chloride for Injection) will be administered IM.
  Arms: Arm B: Placebo for GEO-D03 and MVA/HIV62B

SUMMARY:
The purpose of this study is to evaluate the safety of two HIV vaccines in HIV-1-infected young adults who are taking anti-HIV medications and have very low virus levels. This study will also look at how the immune system responds to the vaccines.

DETAILED DESCRIPTION:
This study will evaluate the safety and immune response of the combination of two vaccines: a multigene DNA HIV-1 vaccine that also expresses GM-CSF (GEO-D03) and a MVA HIV-1 (MVA/HIV62B) vaccine. HIV-1-infected young adults who have suppressed viral levels, have likely acquired (Clade B) HIV-1 infection from sexual contact, and are on highly active antiretroviral therapy (HAART) will be randomly assigned to one of two study arms. Arm A participants will receive the GEO-D03 vaccine at entry and Week 8 and the MVA/HIV62B vaccine at Weeks 16 and 24. Arm B participants will receive placebo vaccines at entry and at Weeks 8, 16, and 24.

Study duration will be 120 weeks (24 weeks for vaccinations plus 96 weeks of follow-up). Study participants will remain on HAART throughout the study. Study visits will occur at screening, entry, and at Weeks 1, 8, 9, 16, 17, 24, 25, 36, 48, 72, 96, and 120. At each study visit, participants will undergo blood collection, a physical exam, and an adherence assessment. At screening, participants will also undergo an electrocardiogram (ECG) and urine collection. Some blood samples will be stored for future use.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected. More details on this criterion can be found in the protocol.
* Likely HIV-1 acquisition in North America or Europe (in the opinion of the site investigator)
* Likely HIV-1 acquisition from sexual transmission (in the opinion of the site investigator)
* On stable HAART, defined as at least three different antiretrovirals (ARVs) from two different classes, with plasma HIV-1 RNA levels fewer than 100 copies/mL for at least 12 months prior to screening. Furthermore, at least two plasma HIV-1 RNA levels fewer than 100 copies/mL (and none with plasma HIV-1 RNA levels 100 or more copies/mL), separated by at least 3 months must have been documented during the 6-month period prior to enrollment.
* Ability and willingness of participant to provide signed written informed consent
* CD4 count 400 cells/mm^3 or greater at screening
* The following lab values (at screening visit):

  * Creatine phosphokinase no higher than 5 times the upper limit of normal (ULN). More details on this criterion can be found in the protocol.
  * Troponin I no more than 1.0 times ULN
  * Hemoglobin greater than 10 g/dL
  * Absolute neutrophil count greater than 1,000 mm^3
  * Platelets greater than 100,000 mm^3
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) no greater than 1.5 times ULN
  * Total bilirubin no greater than 1.5 times ULN (less than 5 times ULN if taking atazanavir)
  * Creatinine less than 2.0 mg/dL
* Female participants who engage in sexual activity that could lead to pregnancy must agree to avoid pregnancy and to consistently use two methods of contraception, including at least one form of barrier contraception, from the screening visit until 90 days after the final vaccination. Medically acceptable contraceptives include barrier methods (such as a condom or diaphragm) used with a spermicide, an intrauterine device (IUD), or approved hormonal contraceptives, such as birth control pills, Depo Provera, or Lupron Depot. Condoms are recommended because their appropriate use is the only contraception method effective for preventing HIV-1 transmission. Two methods of barrier contraception (condom and diaphragm) may be combined to meet this requirement. Sexually active female study participants without reproductive potential are eligible without requiring the use of contraception. Written or oral documentation communicated by clinician or clinician's staff from one of the following is required for participants: physician report/letter or discharge summary.
* To prevent pregnancies, male participants must agree to not attempt to impregnate a female or participate in sperm donation programs. Males engaging in sexual activity that could lead to pregnancy must use a condom from the date of receipt of the first study vaccine until 90 days after receipt of the last study vaccine.
* To prevent HIV-1 transmission to a partner, all participants participating in sexual activity must agree to use effective barrier methods (condoms)
* Willing to comply with all study requirements, including adherence to ARV treatment as prescribed by regular healthcare provider and the expectation to be available for the duration of the study

Exclusion Criteria:

* Documentation of infection with HIV-1 other than Clade B (e.g., if genotype data are available from pre-treatment viral resistance analyses)
* Documentation that the last CD4 T-cell count prior to the initiation of ARV was fewer than 300 cells/mm^3
* Hepatitis B surface antigen positive
* Hepatitis C virus RNA positive
* History of or known active cardiac disease including:

  * evidence of past or evolving myocardial infarction
  * angina pectoris
  * congestive heart failure with permanent sequelae
  * cardiomyopathy (hypertrophic or dilated)
  * myocarditis
  * pericarditis
  * clinically significant arrhythmia (including any arrhythmia requiring medication, treatment, or clinical follow-up)
  * stroke or transient ischemic attack
  * anginal chest pain or shortness of breath with mild activity (such as walking upstairs) due to cardiac disease (New York Heart Association [NYHA] class 2-4)
* Screening ECG with clinically significant findings or features that would interfere with the assessment of myo/pericarditis, including any of the following:

  * Conduction disturbance (complete left or complete right bundle branch block or nonspecific intraventricular conduction disturbance with QRS greater than 120 ms, atrioventricular (AV) block of any degree, or QTc prolongation (greater than 450 ms)
  * Pathologic repolarization (ST segment or T wave) abnormality
  * Significant atrial or ventricular arrhythmia
  * Frequent atrial or ventricular ectopy (e.g., frequent premature atrial contractions, multifocal or two or more premature ventricular contractions in a row)
* Clinically significant, HIV-related renal disease at screening or enrollment (creatinine at least 2.0 mg/dL; persistent high grade proteinuria greater than 2+). If either of these findings is present at screening, tests may be repeated once with option for enrollment if these findings resolve.
* Past or present, HIV-related neurocognitive disease identified by a care provider
* Known hypersensitivity to vaccine components
* Receipt of chemotherapy for active malignancy in the past 12 months
* Prior vaccinations with any HIV-1 vaccine
* Prior immunization with any poxvirus, including vaccinia
* Receipt of immunomodulatory agents, oral or injected systemic corticosteroids for more than 7 days at a time (including nonprescription street steroids), gamma globulin, or investigational agents within 6 months of screening. Use of intranasal or inhaled corticosteroids is allowed.
* Receipt of any other live licensed vaccine within 4 weeks or inactivated licensed vaccine within 2 weeks prior to study enrollment
* Pregnancy or breastfeeding
* Current documented or suspected serious bacterial infection, metabolic illness, malignancy, or immediate life-threatening conditions
* Any clinically significant diseases (other than HIV infection) or clinically significant findings during the screening medical history or physical examination that, in the site investigator's opinion, would compromise the outcome of this study
* Active alcohol or substance abuse (abuse is defined as use of alcohol or other substance such that it is likely to interfere with the ability of the participant to adhere to medications or to return for study visits or is likely to lead to AEs)
* Any foreseeable circumstances that, in the opinion of the site investigator, are likely to jeopardize participant adherence to HAART (i.e., insurance problems, housing instability, or unemployment)

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Grade 3 or higher adverse events (AEs) | Measured through Week 120
Progression of HIV disease status: immunological decline | Measured through Week 120
  Immunological decline defined as a fall in CD4 T-cell count to fewer than 350 cells/mm^3 OR a decline to a level less than 50 percent of baseline, if baseline CD4 T-cell count is more than 700 cells/mm^3 at study entry
Progression of HIV disease status: RNA 1,000 copies/mL or greater measured on two occasions at least 1 week apart | Measured through Week 120
Progression of HIV disease status: development of an AIDS-defining opportunistic infection or malignancy | Measured through Week 120
A greater than or equal to two-fold increase in the frequency of responding HIV-1 Gag-specific CD8 T cells between entry visit and Week 17 visit | Measured through Week 17

SECONDARY OUTCOMES:
Grade 3 or higher AEs at least possibly related to study treatment | Measured through Week 120
A greater than or equal to two-fold increase in the frequency of responding HIV-1 Gag-specific CD8 T cells per individual between entry visit and Week 25 visit | Measured through Week 25

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Greenough, MD, Study Chair — University of MA Medical School (UMMS)-II Biotech

REFERENCES:
- [Background] Rosenberg ES, Graham BS, Chan ES, Bosch RJ, Stocker V, Maenza J, Markowitz M, Little S, Sax PE, Collier AC, Nabel G, Saindon S, Flynn T, Kuritzkes D, Barouch DH; AIDS Clinical Trials Group A5187 Team. Safety and immunogenicity of therapeutic DNA vaccination in individuals treated with antiretroviral therapy during acute/early HIV-1 infection. PLoS One. 2010 May 10;5(5):e10555. doi: 10.1371/journal.pone.0010555. PMID 20479938
- [Background] Persaud D, Luzuriaga K, Ziemniak C, Muresan P, Greenough T, Fenton T, Blackford A, Ferguson K, Neu N, Cunningham CK. Effect of therapeutic HIV recombinant poxvirus vaccines on the size of the resting CD4+ T-cell latent HIV reservoir. AIDS. 2011 Nov 28;25(18):2227-34. doi: 10.1097/QAD.0b013e32834cdaba. PMID 21918423
- [Background] Goepfert PA, Elizaga ML, Sato A, Qin L, Cardinali M, Hay CM, Hural J, DeRosa SC, DeFawe OD, Tomaras GD, Montefiori DC, Xu Y, Lai L, Kalams SA, Baden LR, Frey SE, Blattner WA, Wyatt LS, Moss B, Robinson HL; National Institute of Allergy and Infectious Diseases HIV Vaccine Trials Network. Phase 1 safety and immunogenicity testing of DNA and recombinant modified vaccinia Ankara vaccines expressing HIV-1 virus-like particles. J Infect Dis. 2011 Mar 1;203(5):610-9. doi: 10.1093/infdis/jiq105. Epub 2011 Jan 31. PMID 21282192